CLINICAL TRIAL: NCT05957484
Title: The Clinical and Functional Imaging Effects of Non-invasive Neuromodulation on Illness Awareness in Schizophrenia
Brief Title: The Effects of Non-invasive Neuromodulation on Illness Awareness in Schizophrenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study device no longer available.
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Scion NeuroStim (Industry)
Responsible Party: Principal Investigator, Philip Gerretsen, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 105-2017
Record Dates: First submitted 2023-06-13; First posted 2023-07-24 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia; Anosognosia
Keywords: Non-invasive neuromodulation; Illness awareness; Magnetic resonance imaging; Medical device
MeSH Terms: conditions — Schizophrenia; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Active Treatment (Active Comparator): Study participants will receive ~18-minute active stimulation twice daily over 4 weeks, using a non-invasive brainstem modulation device.
  Interventions: Device: Investigational brainstem neuromodulation device
- Sham Treatment (Placebo Comparator): Study participants will receive ~18-minute of sham stimulation twice daily over 4 weeks using a non-invasive brainstem modulation device.
  Interventions: Device: Investigational brainstem neuromodulation device
- Open Label (Experimental): After completion of sham or active stimulation over 4 weeks, participants can choose to receive ~18-minute active stimulation twice daily for up to 12 weeks.
  Interventions: Device: Investigational brainstem neuromodulation device

INTERVENTIONS:
Device: Investigational brainstem neuromodulation device — This study device is non-invasive meaning it stays outside of the body. It stimulates activity in the brain through a headset with metallic earpieces that fit into the participant's ear canals. The device will be loaded with certain neurostimulation pattern, and the earpieces will provide the stimulation at the prescribed pattern.

SUMMARY:
This study aims to determine the clinical and functional imaging effects of serial CVS on illness awareness in schizophrenia. Specifically, the investigators aim to:

1. Determine if twice-daily CVS for 4 weeks will improve illness awareness compared to the sham condition in participants with schizophrenia. Illness awareness will be assessed at pre- and post-CVS, and weekly thereafter for 4 weeks.
2. Examine changes in brain network activity (blood oxygen level dependent-BOLD in response to an illness awareness task) pre- and post-CVS. This will serve as a biomarker to rigorously test whether repeated CVS engages the PPA associated with illness awareness.

DETAILED DESCRIPTION:
The proposed study employs a novel approach to determine the clinical and functional imaging effects of CVS on illness awareness in schizophrenia - a significant contributor to medication non-adherence and poor treatment outcomes, and arguably the most treatment resistant manifestation of the disorder. CVS is a traditionally safe and non-invasive method of vestibular stimulation that will be used in conjunction with a neuroimaging biomarker to measure brain changes associated with CVS and illness awareness. The results of this study will provide solid evidence for larger treatment-controlled effectiveness studies to determine if CVS is a practical means of producing lasting effects on illness awareness in individuals with schizophrenia or whether maintenance CVS treatment is required.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female inpatients or outpatients ≥ 18 years of age
2. Having a DSM-V diagnosis of schizophrenia or schizoaffective disorder
3. Voluntary and capable of consenting to participation in the research study
4. Fluent in English
5. Moderate-to-severe lack of illness awareness ≤7 on the VAGUS-SR, which corresponds to a rating of ≥3 on PANSS G12 Insight and Judgment item)
6. On a stable dose of antipsychotic and other concomitant medications for at least 2 months, and unlikely to undergo changes in dose during the study

Exclusion Criteria:

1. Unwilling or unable to consent to the study
2. Use of hearing aids or cochlear implants, chronic tinnitus, temporomandibular joint disease
3. Had eye surgery within the previous three (3) months
4. Ear surgery within 6 months prior to entering the study
5. Active ear infection or perforated tympanic membrane
6. Diagnosis of vestibular dysfunction
7. Unstable medical illness or any concomitant major medical or neurological illness, including a history of cardiovascular disease and seizures
8. Acute suicidal and/or homicidal ideation
9. Formal thought disorder rating ≥4 on PANSS item P2
10. DSM-V substance dependence (except caffeine and nicotine) within one month prior to entering the study
11. Positive urine drug screen at the screening visit
12. Metal implants or a pacemaker that would preclude the MRI scan
13. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Illness awareness | Illness awareness will be assessed at pre-intervention and immediately following the intervention and weekly for up to 4 weeks post-intervention.
  Changes in illness awareness will be assessed using questionnaires.

SECONDARY OUTCOMES:
Brain network activity | At baseline and post-intervention.
  Assess changes in brain network activity (blood oxygen level dependent-BOLD in response to an illness awareness task)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gerretsen, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — http://www.camh.net/research